CLINICAL TRIAL: NCT00383630
Title: The Effect of Intramyocardial Injection of Immunoselected Bone Marrow Cells on Myocardial Function in LVAD Bridge to Transplant Patients
Brief Title: Bone Marrow Cell Transplantation to Improve Heart Function in Individuals With End-Stage Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to logistical barriers to cell processing and poor enrollment
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Yoshifumi Naka, Professor of Surgery, Department of Surgery CT, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAC2128; P50HL077096 (NIH); P50HL077096-01 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure, Congestive
Keywords: End Stage Heart Failure; LVAD; Bone Marrow Transplantation; Stem Cell Transplantation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Intramyocardial injection of bone marrow mononuclear cells + LVAD
  Interventions: Biological: Intramyocardial injection of bone marrow mononuclear cells
- Group 2 (Experimental): Intramyocardial injection of CD34+ selected bone marrow mononuclear cells + LVAD
  Interventions: Biological: Intramyocardial injection of CD34+ selected bone marrow mononuclear cells
- Group 3 (Other): LVAD alone
  Interventions: Device: LVAD alone

INTERVENTIONS:
Biological: Intramyocardial injection of bone marrow mononuclear cells — 6mL of bone marrow mononuclear cells will be injected into the myocardium during LVAD implantation.
  Other Names: BMCs + LVAD
  Arms: Group 1
Biological: Intramyocardial injection of CD34+ selected bone marrow mononuclear cells — 6mL of CD34+ selected bone marrow mononuclear cells will be injected into the myocardium during LVAD implantation.
  Other Names: CD34+ selected BMCs + LVAD
  Arms: Group 2
Device: LVAD alone — LVAD implantation without any intramyocardial injection of bone marrow cells.
  Arms: Group 3

SUMMARY:
Heart failure is a condition in which the heart is unable to pump enough blood to the body's other organs. A heart transplant may be necessary for some individuals with end-stage heart failure. Left ventricular assist devices (LVADs) can assist the heart in pumping blood, and are commonly used until a donor heart becomes available. Bone marrow cells injected into the heart may improve heart function and may lead to earlier LVAD removal. The purpose of this study is to evaluate the safety and effectiveness of injected bone marrow cells in improving heart function in individuals with LVADs who are awaiting heart transplants.

DETAILED DESCRIPTION:
Congestive heart failure affects 5 million people in the United States, and over 60,000 are diagnosed with end-stage heart failure. Treatment options for these individuals are extremely limited. Because of a limited supply of donor organs, fewer than 3,000 people receive heart transplants each year. LVADs are battery-operated devices that can act as a temporary solution until a donor heart becomes available. Upon being surgically implanted into a weakened heart, the LVAD mechanically pumps blood from the heart to the rest of the body. There are, however, serious risks associated with LVADs, including infection, blood clots, and stroke. Early removal of the LVAD may be possible by injecting stem cells to regenerate new heart cells and improve heart function. The purpose of this study is to compare the safety and effectiveness of two types of bone marrow cells -- bone marrow mononuclear cells (BMCs) and immunoselected CD34+ hematopoietic stem cells -- in improving heart function in individuals with end-stage heart failure.

This study will enroll individuals undergoing surgery to receive an LVAD. Participants will be randomly assigned to one of following three groups:

Group 1 (n=30): participants will undergo intramyocardial injection of bone marrow mononuclear cells (BMCs) during LVAD implantation

Group 2 (n=30): participants will undergo intramyocardial injection of immunoselected CD34+ hematopoietic stem cells during LVAD implantation

Group 3 (n=15): participants will undergo LVAD implantation

Prior to LVAD implantation, participants in Groups 1 and 2 will have a sample of bone marrow removed. Following LVAD implantation, study visits will occur at Days 45 and 90, and then every 60 days thereafter until participants receive a heart transplant. At each visit, participants will undergo a LVAD wean procedure, during which the mechanical pump of the LVAD will be gradually turned off, and the LVAD will be operated with a hand pump. The length of time that a participant tolerates the wean procedure will be evaluated. Heart size and function, blood flow, and nerve function will also be assessed. Some participants will undergo a 6-minute walk test. At the time of heart transplant surgery, the LVAD will be removed, and heart cell regeneration and heart function will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent, release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documents
* Male, postmenopausal female, or female who may become pregnant but is using adequate contraceptive precautions (defined as use of oral contraceptive, intrauterine devices, surgical contraception, or a combination of a condom and a spermicide), with negative pregnancy test
* Admitted to the clinical center at the time of study entry
* Listed with United Network for Organ Sharing (UNOS) for cardiac transplantation
* Clinical indication and accepted candidate for implantation of an FDA approved LVAD as a bridge to transplantation
* Hemoglobin between 9.0 gm/dl and 16.1 gm/dl within 24 hours prior to study entry
* Platelet count between 100,000/ul and 450,000/ul within 24 hours prior to study entry
* White blood cell count between 2,500/ul and upper limit of normal within 24 hours prior to study entry

Exclusion Criteria

* Cardiothoracic surgery within 30 days prior to study entry
* Myocardial infarction within 6 months prior to study entry
* Prior cardiac transplantation, left ventricular (LV) reduction surgery, or cardiomyoplasty
* Acute reversible cause of heart failure (e.g., myocarditis, profound hypothyroidism)
* Anticipated requirement for biventricular mechanical support
* Stroke within 30 days prior to study entry
* Received investigational intervention within 30 days of study entry
* Pregnant or breastfeeding at time of study entry
* HIV positive within 30 days prior to study entry
* Active systemic infection within 48 hours prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshifumi Naka, MD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - Columbia University, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Subjects: Total number of subjects in the study; breakdown of the number per arm is not available.
Period: Overall Study
Arm/Group | Study Subjects
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Information is not available for the 1 subject.
Arm/Group | Study Subjects
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Time (Minutes) a Patient is Able to Tolerate Wean
Description: This defines the functional status. Due to poor enrollment, data was not analyzed.
Time Frame: Measured 90 days post-intervention
Population: The study was terminated early due to logistical barriers to cell processing and poor enrollment and therefore sufficient data was not obtained for data analysis. Data analysis could not be performed.
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Prevalence of Normal Echocardiographic Assessments
Description: Echocardiographic assessments of myocardial size and function by transthoracic echocardiography with the LVAD at full support, and as tolerated at 1, 5, 10 and 15 minutes following initiation of hand pumping.
  Due to poor enrollment, data was not analyzed.
Time Frame: Measured at baseline, Days 45 and 90 post-intervention, every 60 days thereafter until transplant
Population: as for outcome 1
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Who Completed a Six Minute Walk
Description: 6 Minute walk as tolerated at 15 minutes following initiation of hand pumping.
  Due to poor enrollment, results was not analyzed.
Time Frame: Measured at Days 45 and 90 post-intervention, every 60 days thereafter until transplant
Population: as for outcome 1
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Study Subjects
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Subjects (N=1)
Shock (General disorders) | 1 (1) — Required or Prolonged hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Subjects (N=1)
Renal Dysfunction (General disorders) | 1 (1)
Blood Clot (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes